CLINICAL TRIAL: NCT02331381
Title: A Pilot Study of Imaging and Plan Workflow in a Novel Low-Field Magnetic Resonance Imaging (MRI) Radiotherapy Device
Brief Title: Imaging and Plan Workflow in a Novel Low-Field Magnetic Resonance Imaging (MRI) Radiotherapy Device
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201311081
Record Dates: First submitted 2015-01-02; First posted 2015-01-06 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Cancer; Malignant Tumor
MeSH Terms: conditions — Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- MRI (Experimental): Participants will have a custom immobilization device created for them for the purpose of the study. They will be scanned from one to four occasions during radiation treatment. If enrolled in the study prior to the first radiation treatment, the first imaging scan may be scheduled prior to the first radiation treatment, with subsequent scans during treatment separated by at least one day. Patients will be in the scanner for approximately 30 minutes to one hour, either prior to or following their standard of care radiotherapy treatment.
  Interventions: Device: Magnetic resonance imaging

INTERVENTIONS:
Device: Magnetic resonance imaging
  Other Names: MRI

SUMMARY:
The results of this imaging and treatment planning protocol will aid in developing procedures for patient localization and future clinical implementation of low-field MRI to confirm positioning prior to radiation treatment. Images acquired during this study may aid future study design for adaptive planning based on low-field MRI images. Moreover, results of this imaging and treatment planning may lead to guidance on optimal use of this novel device.

DETAILED DESCRIPTION:
Recently, Viewray Inc (Cleveland, OH) has released the RenaissanceTM System 1000, which consists of the combination of an open, split solenoid 0.35 T MRI scanner that is equipped for parallel imaging with a 60Co gamma-ray radiation treatment unit. The MRI scanner is required to be a low field unit to allow for imaging with spatial integrity by limiting magnetic susceptibility artifacts due to the patient and to prevent significant perturbations of the dose distribution. The 0.35 T magnet is a variant of the Siemens MAGNETOM product used for intraoperative imaging.

A previous study of pilot imaging using this device without the 60Co sources was completed in 2012 (HRPO# 201105295). In this study, a total of 26 patients were imaged with the device. Fourteen of these patients also had onboard CT imaging (OB-CT) where the two sets of imaging and relative organs at risk (OARs) could be compared. Fifteen to 24 OARs were evaluated per anatomical site. In total, 221 OARs and 10 target structures were compared for visualization on MRI and OB-CT image sets by each physician. At least 2/3 physicians evaluated MRI as offering better visualization for 71% of structures, OB-CT offering better visualization for 10% of structures, and both offering equivalent visualization for 14% of structures. Physicians agreed unanimously for 74% and in majority for >99% of structures evaluated, respectively. For <1% of structures, no consensus was reached. Targets were better visualized on MRI in 4/10 cases, and were never better visualized on OB-CT images.

There were limitations to this prior study. The patients were not imaged in immobilization devices that are commonly used in radiation therapy. This precluded the creation of a mock radiation therapy plan using the device for these patients. Also, the device was not evaluated in the context of radiation therapy decision making, such as patient shifts, target localization and patient repositioning.

The purpose of this study is to evaluate the imaging and plan workflow for radiation therapy utilizing this novel device. For this protocol, only the MRI scanner of the machine will be utilized. The 60Co portion of the machine capable of radiation treatment administration will not be utilized, and there will be no experimental treatments or modifications to each patient's standard of care radiation treatment plan.

ELIGIBILITY:
Eligibility Criteria:

* Scheduled to receive radiation therapy.
* At least 18 years of age.
* Does not meet any standard contraindications for MRI (such as being claustrophobic, having metal objects within the body that cannot be removed or having large tattoos), confirmed by completion of our clinical MRI questionnaire form
* Able to understand and willing to sign an IRB approved written informed consent document.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-12-26 (Actual); Primary Completion 2015-12-23 (Actual); Study Completion 2016-09-07 (Actual)

PRIMARY OUTCOMES:
Adequacy of the radiation therapy plan | Duration of radiation therapy
  The radiation plan will be evaluated based on the recorded clinical goals prescribed by the attending physician. Plans will be classified as 'adequate' if they meet the prescribed goals for the clinical radiation therapy plan.
Feasibility of patient localization workflow | Duration of radiation therapy
  The localization time will be classified as 'adequate' if it is less than or equal to 15 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Michalski, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu